CLINICAL TRIAL: NCT06324760
Title: Usefulness of Alpha-lipoic Acid Combined With B Vitamins for the Treatment of Restless Legs Syndrome
Brief Title: Alpha-lipoic Acid Combined With B Vitamins Shows Promise for Treating Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: Uriach Consumer Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: LIPOICSPI2018
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Restless Legs Syndrome
Keywords: RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Vitamin B Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Dietary Supplement: Alpha-lipoic acid combined with B vitamins — The investigational product utilized in this research, Tiobec® 400 is a dietary supplement enriched with ALA, B vitamins, and vitamins E and C. T400 is designed to mitigate oxidative stress and support the optimal functioning of the nervous system

SUMMARY:
Investigating Tiobec® 400's efficacy in alleviating Restless Legs Syndrome symptoms sheds light on promising therapeutic avenues.

DETAILED DESCRIPTION:
Restless legs syndrome, also known as Willis-Ekbom disease, is a neurological disorder characterised by uncomfortable sensations in the legs and an urge to move them. In Spain, its prevalence range is estimated to be between 11.6% - 19.5% in adults, but it is difficult to know due to underdiagnosis. Alpha-lipoic acid (ALA) and B vitamins have emerged as potential treatments due to their roles in reducing oxidative stress and associated vitamin deficiencies. The Tiobec® 400 (T400) supplement combines ALA, B vitamins, E, and C, and its efficacy and safety in alleviating RLS symptoms, along with its impact on anthropometric measures, are under investigation. This study aims to explore therapeutic options for managing RLS, with promising results.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a minimum of 18 years of age.
* They must have a primary diagnosis of RLS without prior therapeutic interventions for the ailment.
* They need to provide explicit consent via an informed consent document.

Exclusion Criteria:

* Patients diagnosed with pathologies other than RLS that affect sleep quality.
* Those with persistent renal diseases or any other chronic, severe medical condition.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data will be collected from patients who meet the selection criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Measure the subjective RLS symptoms of the participants through the IRLSSG rating scale (IRLS) | 6 months
  This scale contains 10 items, rated from 0 to 4, according to the severity reported by the patient (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.). The cumulative scores are categorized as mild (1-10), moderate (11-20), severe (21-30), and very severe (31-40).

SECONDARY OUTCOMES:
Anthropometric parameters of the patients. | 6 Months
  Weight (kg).
Patients' body measurements | 6 Months
  Body mass index (BMI) (kg/m²).
Measurements of patient anatomy | 6 Months
  Total fat mass (kg).
Patients' body characteristics. | 6 Months
  Visceral fat mass (kg).
Measurements of patient anatomy. | 6 Months
  Muscle mass (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Albares, Doctor, Principal Investigator — Centro Medico Teknon
Locations (1):
- Medical Center Teknon, Barcelona, Spain